CLINICAL TRIAL: NCT03955523
Title: Effects of a Single Exercise Session or Meal on Physical and Mental Health of People With Spinal Cord Injury: a Case Series Study
Brief Title: Single Exercise Session or Meal vs Control in SCI: Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kathleen Martin Ginis, professor, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Case series exercise/meal SCI
Record Dates: First submitted 2019-05-14; First posted 2019-05-20 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injuries
Keywords: SCI; paraplegia; tetraplegia; quadriplegia; spinal cord
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Intervention Model Description: Case series: intraindividual analyses comparing single exercise trial vs single diet trial vs control (doing nothing)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single exercise bout trial (Experimental): Exercise trial day: 30 min of continuous exercise at 60% VOpeak (or at the least 3 bouts of 10 min at 60% VO2peak separated by no more than 1 minute rest) - power output is set at that determined during the maximum test on the first visit, and adjusted accordingly if there is a deviation >5% VO2peak for at least 3 minutes of exercise.
  Interventions: Other: Single exercise bout trial
- Single diet trial (Experimental): Diet trial day The protocol of the diet trial day is identical to that of the exercise trial day, except that exercise is substituted by asking the participant to eat a standardized breakfast meal that it is commonly consumed in a fast-food chain (i.e. cheese and egg McMuffin, double portion of hash browns and an orange pop).
  Interventions: Dietary Supplement: Single diet trial
- Control (doing nothing) (No Intervention): Non-exercise trial day The protocol of the non-exercise trial day is identical to that of the exercise trial day, except that exercise is substituted by 30 min of quiet sitting in a lounge area (e.g. reading, working or watching a movie on an electronic device) without further engagement with other people.

INTERVENTIONS:
Other: Single exercise bout trial — Exercise trial day: 30 min of continuous exercise at 60% VOpeak (or at the least 3 bouts of 10 min at 60% VO2peak separated by no more than 1 minute rest) - power output is set at that determined during the maximum test on the first visit, and adjusted accordingly if there is a deviation >5% VO2peak for at least 3 minutes of exercise.
  Arms: Single exercise bout trial
Dietary Supplement: Single diet trial — Diet trial day The protocol of the diet trial day is identical to that of the exercise trial day, except that exercise is substituted by asking the participant to eat a standardized breakfast meal that it is commonly consumed in a fast-food chain (i.e. cheese and egg McMuffin, double portion of hash browns and an orange pop).
  Arms: Single diet trial

SUMMARY:
The purpose of this study is to examine the immediate effects of a single exercise session or a high fat/high carbohydrate meal on the physical and mental health of people with a spinal cord injury (SCI). Specifically, we want to better understand the responses in people with SCI when they conduct exercise or eat an unhealthy meal, when looking at inflammation levels, the number and function of immune cells, brain function, pain and how one feels (affect). If we can understand these responses, then clinicians, sports practitioners and dieticians can provide better advice to people with SCI.

DETAILED DESCRIPTION:
Background / justification Exercise training and diet interventions can influence the chronic low-grade inflammatory state common among people with SCI. However, little is known about mechanisms underlying such changes. In SCI, changes in cytokines reflecting an inflammatory state are observed after long-term exercise training and diet interventions. After a single exercise bout, mixed results in cytokine responses have been observed, while the effects of a single meal on cytokines responses have never been studied in SCI. As indicated by research in other clinical populations, changes in immune cell count and immunephenotyping may precede and underlie changes in an inflammatory state. Given immunological changes post-SCI, this hypothesis needs to be tested in people with SCI.

Similarly, very little is known about exercise-induced changes in cognitive function in people with SCI, despite the improvements found in other clinical populations. One mechanism potentially underlying the effects of exercise on cognition, is an increase in brain-derived neurotrophic factor (BDNF), which has been observed in able-bodied people after a single bout of exercise Given cerebrovascular changes and potential cognitive dysfunction post-SCI this hypothesis needs to be tested in people with SCI.

Exercise training has also been identified as a potential strategy for improving mental health in adults with SCI who on average report poorer mental health than adults without disabilities However, little is known about mechanisms underlying positive effects of exercise on mental health of people with SCI. It is not clear whether a single standardised exercise bout immediately leads to improvements in affect and perceived stress, and if positive effects of a single exercise bout are mediated by reductions in neuropathic pain Additionally, exercise has been reported to be effective in the alleviation of other types of pain commonly experienced by people with SCI, for example musculoskeletal (MSK) pain. Conducting an exercise intervention in accordance with validated international SCI exercise guidelines for improving cardiometabolic health will not only allow us to determine the effects of the guidelines on MSK and NP pain, but also identify potential mechanisms by which exercise reduces pain.

Taken together, SCI pilot data is needed to gain support for the inclusion of the above-described outcomes in long-term exercise training or diet intervention studies (e.g. RCTs). Such evidence is needed to understand how exercise training and diet interventions for people with SCI can be maximally effective. Ultimately, this will allow clinicians, sports practitioners and dieticians to provide better advice to people with SCI, and provide people with SCI with the opportunity to make evidence-based health choices.

Purpose and objectives

The purpose of this pilot study is to examine the immediate effects of a single exercise session or a typical unhealthy meal on inflammation, immune cell count/phenotyping, brain function, pain, affect and perceived stress in people with SCI. Specific objectives are to compare the effects of a 30-min upper-body arm crank exercise session at 60% peak oxygen uptake or a high fat/high carbohydrate meal from a fast-food chain to a control condition in which participants sit quietly for 30 minutes. Outcomes selected will be:

* inflammation (measurement and function of cytokines IL-6, IL-10 and TNF-alpha)
* immune cell count/phenotyping (cell numbers per ml blood and percentage total leukocytes for monocytes, neutrophils, eosinophils, T cells, B cells and natural killer cells)
* brain function (task-switching test, Stroop test and BDNF]
* neuropathic pain (Neuropathic Pain Scale distinguishing 10 neuropathic pain qualities)
* - Musculoskeletal pain (Musculoskeletal Pain Scale measuring 2 dimensions of musculoskeletal pain qualities)
* affect (Feeling Scale and Felt Arousal Scale)

Research design Given the novelty of this topic and pilot nature of this study, a case series study design is most appropriate: it will reduce the burden and cost of recruiting a relatively large group of people with SCI, while maximizing insight into intra-individual responses [Published case series of individuals with SCI typically include 5--10 cases This case series study will include 4 research visits on 4 separate days taking place across two weeks with a minimum of 48 h between days. After receiving the written informed consent via email or mail (see the sections on recruitment and obtaining consent below), the participant will be invited for the first visit: a screening/familiarisation visit. This first visit is followed by (in randomized order): an exercise trial day, a diet trial day and a control trial day. Further details on inclusion criteria, exclusion criteria, recruitment and study procedures are provided in the sections below.

Statistical analysis Group descriptives (median, interquartile range, mean, standard deviation) will be calculated for all participant characteristics, outcome measures at the different time points, and the absolute and relative change in outcomes measures across the different time points.

Data will be further analyzed at both the group level and the individual level. At the group level, ANOVA or non-parametric equivalent (subject to the distribution of the data) will be conducted to test whether outcomes change across the different time points and whether these changes are different from those observed in the control condition. At the individual level, data will be plotted for each participant to examine changes across the different time points on each trial day. Where necessary, further insight into individual patterns is gained by visualizing data

ELIGIBILITY:
Inclusion Criteria:

* Published case series of individuals with spinal cord injury (SCI) typically include 5-10 cases (Todd & Martin Ginis, 2018).

For this study, we aim to include 7 individuals who are provincial wheelchair rugby players or individuals who train for an equivalently high-intensity sport (e.g. wheelchair racing, hand cycle racing, para alpine skiing) - all participants should be performing training at least 3 times per week at a high-intensity. Men and women are recruited through community partners in the Okanagan region, if aged 18+, with chronic spinal cord injury (longer than 1 year post-injury), injury levels at the third cervical level or below (as long as diaphragmatic control and arm functioning allow upper-body exercise), American Spinal Cord Injury Association Impairment Scale classifications A-D, upper-arm veins accommodating 3 venepunctures per day, the ability to read and write in English, and no contraindications to maximal exercise based on the latest guidelines of the American College of Sports Medicine (2013).

These individuals are sampled to ensure participants are accustomed and acclimated to exercise (both the peak aerobic exercise test and the 30 min of exercise at 60% VO2peak (i.e. moderate to vigorous intensity).

Exclusion Criteria:

* Excluded are people with SCI who do not meet the inclusion criteria and/or:
* are not able to refrain from anti-inflammatory medication (e.g. Ibuprofen, Naproxen, Tylenol) for at least 24h before each trial day
* have a clinically diagnosed metabolic disorder (e.g. diabetes, hypothyroidism), progressive disease (e.g. multiple sclerosis) or mental disorder (e.g. depression)
* are pregnant

Responses of these individuals are not considered to represent those that can be expected in the general population with spinal cord injury (SCI), which is the population that this study is targeting.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Cytokine profile | Before, immediately after and 2 hours post-baseline
  Plasma cytokines (IL6, IL10, TNFalpha) will be measured in plasma by Milliplex® high-sensitivity assay on a MagPIX® multiplex reader.
Immunephenotyping profile | Before, immediately after and 2 hours post-baseline
  Immediately after taking the venous blood sample, immune cell counts will be quantified using the 8-Color Immunophenotyping Kit (130-120-640, Miltenyi Biotec) on a MACSQuant Analyzer 10 Flow Cytometer (Miltenyi Biotec) [3, 4]. Cell numbers per ml blood and percentage total leukocytes for monocytes, neutrophils, eosinophils, T cells, B cells and natural killer cells will be assessed to determine the impact of exercise on the major circulating leukocyte populations.
BDNF | Before, immediately after and 2 hours post-baseline
  Plasma samples will be collected in 3mL EDTA blood tubes and serum will be collected in 3mL serum separator tubes. Samples will be analyzed using a commercially available enzyme-linked immunosorbent assay in accordance with the manufacturer's instructions (Quantikine DBD00 BDNF ELISA, RnD Systems)
Cognitive Function | Before, immediately after and 2 hours post-baseline
  Cognitive function will be assessed using a battery of 2 psychometrically valid tests (task-switching test and Stroop test) administered via a tablet-based app (BrainBaseline, Digital Artefacts). These tests measure selective attention, inhibitory control, and processing speed and will be used given their sensitivity to improvement following an acute bout of exercise [6]. Each test will take less than 3 minutes to complete. There is no prognostic validity to these tests (i.e., assessing cognitive impairment), rather they are intended to demonstrate within- and between-subject changes for research purposes. There are no risks associated with this measure.
Neuropathic pain | Before, immediately after and 2 hours post-baseline
  Neuropathic pain scale, with one question adapted in accordance with repeated measurements of neuropathic pain.
Musculoskeletal pain. | Before, immediately after and 2 hours post-baseline
  Musculoskeletal pain will be measured with a momentary pain intensity scale (2-item, 10 point scale) that has been adapted to be specific for Musculoskeletal pain.
Affect | Before, immediately after and 2 hours post-baseline
  Felt Arousal Scale (6-point, single item scale) and Feeling Scale (11-point, single item scale measures participants' overall feeling of pleasure-displeasure, i.e. -5 = very bad, +5 = very good)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Martin Ginis, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Given the case series design, data is too easy to lead back to individual participants, hence data is not shared.

REFERENCES:
- [Background] Todd KR, Martin Ginis KA. An examination of diurnal variations in neuropathic pain and affect, on exercise and non-exercise days, in adults with spinal cord injury. Spinal Cord Ser Cases. 2018 Oct 27;4:94. doi: 10.1038/s41394-018-0130-3. eCollection 2018. PMID 30393565
- [Background] Barry JC, Simtchouk S, Durrer C, Jung ME, Little JP. Short-Term Exercise Training Alters Leukocyte Chemokine Receptors in Obese Adults. Med Sci Sports Exerc. 2017 Aug;49(8):1631-1640. doi: 10.1249/MSS.0000000000001261. PMID 28319586
- [Background] Post MW, van Leeuwen CM. Psychosocial issues in spinal cord injury: a review. Spinal Cord. 2012 May;50(5):382-9. doi: 10.1038/sc.2011.182. Epub 2012 Jan 24. PMID 22270190
- [Background] Dinoff A, Herrmann N, Swardfager W, Lanctot KL. The effect of acute exercise on blood concentrations of brain-derived neurotrophic factor in healthy adults: a meta-analysis. Eur J Neurosci. 2017 Jul;46(1):1635-1646. doi: 10.1111/ejn.13603. Epub 2017 Jun 19. PMID 28493624
- [Background] Allison DJ, Beaudry KM, Thomas AM, Josse AR, Ditor DS. Changes in nutrient intake and inflammation following an anti-inflammatory diet in spinal cord injury. J Spinal Cord Med. 2019 Nov;42(6):768-777. doi: 10.1080/10790268.2018.1519996. Epub 2018 Oct 2. PMID 30277850
- [Derived] Todd KR, Van Der Scheer JW, Walsh JJ, Jackson GS, Dix GU, Little JP, Kramer JLK, Martin Ginis KA. The Impact of Sub-maximal Exercise on Neuropathic Pain, Inflammation, and Affect Among Adults With Spinal Cord Injury: A Pilot Study. Front Rehabil Sci. 2021 Oct 26;2:700780. doi: 10.3389/fresc.2021.700780. eCollection 2021. PMID 36188763